CLINICAL TRIAL: NCT06923579
Title: Treatment Of Meta-diaphyseal Bone Defect In Long Bone With Titanium Mesh Cage : Case Series Study
Brief Title: Treatment Of Meta-diaphyseal Bone Defect In Long Bone With Titanium Mesh Cage
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Adel Ragab Mohamed, Assissant lecturer, Assiut University
Other Study IDs: Meta-diaphyseal Bone Defect
Record Dates: First submitted 2025-03-25; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Meta-diaphyseal Bone Defect In Long Bone
Keywords: Meta-diaphyseal Bone Defect In Long Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adult patients 16 - 60 years old in both gender
  Interventions: Procedure: Titanium Mesh Cage

INTERVENTIONS:
Procedure: Titanium Mesh Cage — the Harms cage was adapted for long bone reconstruction due to its structural stability and biocompatibility. The cage provides immediate mechanical support while allowing for bone ingrowth, addressing the limitations of traditional methods.
  Advantages of the titanium mesh cage include its ability to maintain bone length, provide immediate stability, and allow for earlier weight-bearing. The porous structure facilitates vascularization and bone integration, potentially leading to improved healing outcomes

SUMMARY:
Meta-diaphyseal bone defects in long bones pose a significant challenge in orthopedic surgery. Traditional treatment methods include autologous bone grafts, allografts, and distraction osteogenesis. Autologous bone grafting is often considered the gold standard due to its superior biological compatibility, but it is limited by complications such as donor site morbidity and the finite quantity of available graft material. Allografts provide an alternative but are associated with risks of immune rejection and disease transmission. Distraction osteogenesis, popularized by Ilizarov, allows for gradual bone regeneration and lengthening but requires prolonged treatment periods and carries the risk of complications like pin tract infections.

In the late 1990s, titanium mesh cages, particularly the Harms cage, emerged as a novel solution for meta-diaphyseal bone defects. Originally developed for spinal surgery, these cages were adapted for long bone reconstruction due to their structural stability and biocompatibility. The cylindrical design of titanium mesh cages provides mechanical support while allowing for the containment of bone graft material and promoting vascular ingrowth. This technique enables effective reconstruction of segmental defects by combining the cage with cancellous bone grafts or other substitutes.

Recent studies have demonstrated promising outcomes with titanium mesh cages in treating meta-diaphyseal defects. High union rates and favorable functional results have been reported in long-term follow-ups. The method offers advantages such as immediate structural stability and adaptability to various clinical scenarios, making it a valuable option for addressing complex bone defects. However, like all techniques, it is not without limitations, including potential complications such as residual limb length discrepancies or recurrent infections in some cases. Nonetheless, titanium mesh cages represent a significant advancement in the management of challenging long bone defects.

DETAILED DESCRIPTION:
Meta-diaphyseal bone defects in long bones present a significant challenge in orthopedic surgery. Traditional treatment methods include autologous bone grafts, allografts, and distraction osteogenesis. Autologous bone grafting, considered the gold standard, is limited by donor site morbidity and the finite availability of graft material. Allografts provide an alternative but carry risks such as immune rejection and disease transmission. Distraction osteogenesis, popularized by Ilizarov, allows for gradual bone lengthening but requires prolonged treatment periods and may lead to complications like pin tract infections. More recently, bioengineered materials and growth factors have been explored as potential solutions, but their clinical application remains challenging.

Open fractures are classified based on orthogonal radiographs to assess the extent and geometry of bone loss. These classifications include incomplete defects (D1), minor or subcritical complete defects (D2), and segmental or critical-sized defects (D3). Incomplete defects (D1) are further divided into D1A (<25% cortical loss), D1B (25-75% cortical loss), and D1C (>75% cortical loss). Minor/subcritical defects (D2) are categorized as D2A (two oblique ends allowing overlap), D2B (one oblique end and one transverse end), and D2C (two transverse ends). Segmental/critical-sized defects (D3) are classified into D3A (moderate defects, 2 to <4 cm), D3B (major defects, 4 to <8 cm), and D3C (massive defects, ≥8 cm). The reliability of these classifications has been assessed using Fleiss' kappa tests among independent observers.

The use of titanium mesh cages, particularly the Harms cage, emerged in the late 1990s as a novel approach for treating meta-diaphyseal bone defects. Initially developed for spinal surgery, the Harms cage was adapted for long bone reconstruction due to its structural stability and biocompatibility. These cages provide immediate mechanical support while promoting bone ingrowth, addressing many limitations of traditional methods. The porous structure facilitates vascularization and integration with surrounding bone, potentially leading to improved healing outcomes.

Titanium mesh cages offer several advantages in managing meta-diaphyseal defects. They maintain bone length, provide immediate stability, and allow for earlier weight-bearing. However, challenges such as the risk of subsidence and the need for precise surgical technique remain. Recent studies have reported high union rates and favorable functional outcomes in long-term follow-ups, suggesting that titanium mesh cages are a reliable option for treating complex long bone defects.

This case series study aims to evaluate the efficacy of titanium mesh cages in addressing meta-diaphyseal bone defects. It focuses on clinical outcomes, radiographic healing, and patient-reported functional improvements. By validating this technique, titanium mesh cages could potentially set a new standard in managing challenging bone defects in orthopedic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age: Patients aged 16-60 years (adults of any gender)
* Defect Location: Meta-diaphyseal defects in long bones (femur, tibia, humerus)
* Defect Size: Critical-sized defects ≥2 cm in length
* Case Type: Both acute (traumatic/post-traumatic) and chronic (osteomyelitis, non-union) presentations
* Exclusion Criteria:
* Soft Tissue Status: Inadequate soft tissue coverage requiring complex reconstruction (unreconstructable defects)
* Infection: Active local or systemic infection (e.g., unresolved osteomyelitis, sepsis)
* Host Status: Severe immunocompromise or systemic conditions contraindicating surgery (e.g., uncontrolled diabetes, renal failure)
* Prior Interventions: Previous failed reconstruction attempts with persistent instability

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients at Assiut university hospitals, Department of Orthopaedics and Traumatology
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-04-10 (Estimated); Primary Completion 2028-03-25 (Estimated); Study Completion 2028-03-25 (Estimated)

PRIMARY OUTCOMES:
Radiographic Bone Union Assessment in Critical-Sized Defects | 1 month
  This primary outcome measure evaluates bone union in critical-sized defects using standardized anteroposterior and lateral X-ray assessments. Union is defined by three key radiographic criteria:
  Bridging trabeculae, Callus maturation and Fracture line resolution

SECONDARY OUTCOMES:
Incidence and rate of complications (e.g. non-union, post-operative infections.....) | 3 months
  This measure evaluates complication rates following titanium mesh cage (TMC) reconstruction for meta-diaphyseal defects. Complications are categorized as:
  Non-union Postoperative infections Hardware-related issues Limb dysfunction

REFERENCES:
- [Background] Feltri P, Solaro L, Di Martino A, Candrian C, Errani C, Filardo G. Union, complication, reintervention and failure rates of surgical techniques for large diaphyseal defects: a systematic review and meta-analysis. Sci Rep. 2022 Jun 1;12(1):9098. doi: 10.1038/s41598-022-12140-5. PMID 35650218
- [Background] Attias N, Thabet AM, Prabhakar G, Dollahite JA, Gehlert RJ, DeCoster TA. Management of extra-articular segmental defects in long bone using a titanium mesh cage as an adjunct to other methods of fixation: a multicentre report of 17 cases. Bone Joint J. 2018 May 1;100-B(5):646-651. doi: 10.1302/0301-620X.100B5.BJJ-2017-0817.R2. PMID 29701099
- [Background] Klezl Z, Bagley CA, Bookland MJ, Wolinsky JP, Rezek Z, Gokaslan ZL. Harms titanium mesh cage fracture. Eur Spine J. 2007 Dec;16 Suppl 3(Suppl 3):306-10. doi: 10.1007/s00586-007-0377-z. Epub 2007 May 12. PMID 17497187
- [Background] Cobos JA, Lindsey RW, Gugala Z. The cylindrical titanium mesh cage for treatment of a long bone segmental defect: description of a new technique and report of two cases. J Orthop Trauma. 2000 Jan;14(1):54-9. doi: 10.1097/00005131-200001000-00011. PMID 10630804
- [Background] Solomon LB, Callary SA, Boopalan PR, Chakrabarty A, Costi JJ, Howie DW. Impaction bone grafting of segmental bone defects in femoral non-unions. Acta Orthop Belg. 2013 Feb;79(1):64-70. PMID 23547518
- [Background] Einhorn TA, Gerstenfeld LC. Fracture healing: mechanisms and interventions. Nat Rev Rheumatol. 2015 Jan;11(1):45-54. doi: 10.1038/nrrheum.2014.164. Epub 2014 Sep 30. PMID 25266456
- [Background] Rosslenbroich SB, Oh CW, Kern T, Mukhopadhaya J, Raschke MJ, Kneser U, Krettek C. Current Management of Diaphyseal Long Bone Defects-A Multidisciplinary and International Perspective. J Clin Med. 2023 Sep 29;12(19):6283. doi: 10.3390/jcm12196283. PMID 37834927
- [Background] Tetsworth KD, Burnand HG, Hohmann E, Glatt V. Classification of Bone Defects: An Extension of the Orthopaedic Trauma Association Open Fracture Classification. J Orthop Trauma. 2021 Feb 1;35(2):71-76. doi: 10.1097/BOT.0000000000001896. PMID 32639397